CLINICAL TRIAL: NCT01831284
Title: Correlates and Consequences of Increased Immune Activation in Injection Drug Users
Status: Completed | Type: Observational
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Other Study IDs: MMA-0774
Record Dates: First submitted 2013-02-28; First posted 2013-04-15 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Intravenous Drug Usage
MeSH Terms: interventions — Sigmoidoscopy; Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sigmoidoscopy with biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- heroin injecting drug users: Sigmoidoscopy with biopsy, in medically stable active injecting drug users
  Interventions: Procedure: Sigmoidoscopy with biopsy
- healthy controls: Sigmoidoscopy with biopsy, in non-injecting controls-
  Interventions: Procedure: Sigmoidoscopy with biopsy
- Former heroin injection drug users: Sigmoidoscopy with biopsy, in former injectors of heroin with or without other agents
  Interventions: Procedure: Sigmoidoscopy with biopsy

INTERVENTIONS:
Procedure: Sigmoidoscopy with biopsy — Sigmoidoscopy with biopsy

SUMMARY:
The goal of this study is to learn how injection drug use may affect the immune system.

DETAILED DESCRIPTION:
The goal of this study is to learn how injection drug use may affect the immune system. One way to measure this is by looking at the blood and the gut, or gastrointestinal tract at the same time. It is thought that activating the immune system by injection drug use may increase destruction of immune cells in the gut. To test this theory, the investigators are enrolling HIV-negative injection drug users, HIV-negative people who do not use drugs and HIV-negative former injection drug users.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Between the ages of 18 and 55
* Absence of medical conditions that would preclude flexible sigmoidoscopy
* Absence of active opportunistic infection requiring active therapy including antibiotics or anti-neoplastics (note this does not include prophylactic antibiotic therapy)

Exclusion Criteria:

* History of bleeding disorder
* Platelet count below 70,000
* INR>1.5 or PTT>2X control
* Active use of anticoagulants or aspirin therapy that cannot be interrupted
* Comorbid diagnosis of inflammatory bowel disease
* Pregnancy, incarceration, mentally disabled individuals
* HIV-1 infection
* Currently on Hepatitis C treatment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Group 1: HIV-uninfected, active IDU defined as a minimum of 3 injections of heroin per week (N=48)
  Group 2: Non-injecting controls defined as no lifetime use of injection drugs and no illicit non-injection opiate or cocaine for at least 3 years (N=48)
  Group 3: Former injectors of heroin with/without other agents will be recruited and followed after approximately 1 month (N=48) and 3 months (N=48) from the time of last injection.
  All groups will be matched for age, sex, and race/ethnicity. Groups 1 and 3 will be matched for Hepatitis C status and HCV RNA levels. Group 1 subjects will be studied twice; at baseline, at 1-2 months to assess stability of findings. Group 2 will be studied once; Group 3 will be studied at 1 and 3 months after ceasing injections.
Sampling Method: Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2012-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Examine the behavioral and immunological correlates of increased immune activation in active and former injection drug users (IDUs) in blood and tissue. | 3 months
  Detailed assessments of blood and GI tissue including measurements of HCV viremia in 1) active HIV-1-uninfected IDUs (N=48) 2) a cohort of individuals entering or in drug treatment programs who have stopped injecting for approximately 1 and 3 months (N=48), the majority of whom we anticipate will be infected with HCV; and 3) non-injecting controls (N=48). In addition to obtaining blood and tissue, we will collect behavioral data including injection and other drug use and sexual behaviors.

SECONDARY OUTCOMES:
Determine the mechanisms of increased immune activation associated with active IDU using a systems biology approach. | 3 months
  This study will isolate specific cell populations from the peripheral blood as well as the GALT that mediate innate and adaptive immune responses. We will perform transcriptional profiling with the goal of identifying gene expression patterns of a-priori defined biological pathways and functional categories that associate with phenotypes of interest. Finally to complement and clarify the results of our in vivo studies, we will examine the in vitro effects of adding morphine and methadone and withdrawing opiates on T cell subsets of interest using a systems biology approach.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Markowitz, MD, Principal Investigator — Aaron Diamond AIDS Research Center
Locations (1):
- The Rockfeller University, New York, New York, United States

REFERENCES:
- [Derived] Markowitz M, Deren S, Cleland C, La Mar M, Silva E, Batista P, St Bernard L, Gettie N, Rodriguez K, Evering TH, Lee H, Mehandru S. Chronic Hepatitis C Virus Infection and the Proinflammatory Effects of Injection Drug Use. J Infect Dis. 2016 Nov 1;214(9):1376-1382. doi: 10.1093/infdis/jiw373. Epub 2016 Aug 11. PMID 27521361